CLINICAL TRIAL: NCT06372587
Title: Leveraging Genetically Encoded engiNeered protEins foR Next-Generation alzheImer'S Therapeutics
Brief Title: Next-Generation alzheImer'S Therapeutics
Acronym: ENERGISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5502
Record Dates: First submitted 2024-04-04; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alzheimer's disease patients (Experimental): To test engineered proteins in human neurons derived from skin biopsy from Alzheimer's disease patients
  Interventions: Other: genetically encoded engineered proteins
- Neurotypical control patients (Sham Comparator): To test engineered proteins in human neurons derived from skin biopsy from neurotypical control patients
  Interventions: Other: genetically encoded engineered proteins

INTERVENTIONS:
Other: genetically encoded engineered proteins — using genetically encoded engineered proteins to obtain an inducible control of their activity in living human neurons promoting synaptic plasticity and/or preventing dendritic spines loss

SUMMARY:
Is this the right time to use next-generation approaches in Alzheimer's disease (AD)? In recent years, several large clinical trials testing treatments for AD have failed, putting the entire field on a reset. AD drug trials have almost exclusively sought to use antibodies targeted toward misfolded amyloid and tau proteins. Of note, although these approaches have failed, they were designed to cover both familial and sporadic forms of AD. On the other hand, the failure in developing new effective drugs is attributed to, but not limited to, the highly heterogeneous nature of AD with multiple underlying hypotheses and multifactorial pathology. The idea underlying this project is based on the assumption that learning and memory disorders can arise when the connections between neurons do not change appropriately in response to experience. Thus, by intervening on the core mechanisms of the cellular correlate of learning and memory, i.e., synaptic plasticity, the investigators expect to preserve some of the essential brain functions in AD. By overcoming the limits of traditional AD therapeutic approaches, the investigators will use genetically encoded engineered proteins (GEEPs), which the investigators developed and tested in vitro and in murine models, to control their activity in living human neurons boosting synaptic plasticity. Indeed, outstanding and relevant progress in understanding synaptic physiology empowers the possibility to prevent or limit brain disease like never before. The investigators designed GEEPs to address some of the leading causes of synaptic plasticity failures documented in AD. Thus, GEEPs will be tested in human induced pluripotent stem cells (hiPSCs)-derived living neurons obtained from reprogrammed peripheral tissues of participants with Alzheimer's diseases. hiPSCs will be obtained from fibroblast-derived from a skin biopsy of participants with AD and controls performed in local anesthesia using a 4 mm punch. The findings will provide the first preclinical study on the effect of genetically engineered proteins to control essential pathways implicated in synaptic plasticity on AD-related cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Manifest clinical criteria for probable AD;
* Age between 18 and 80 years;
* Signed informed consent obtained;

Exclusion Criteria:

* Patients suffering from other neurological diseases;
* Patients with coagulation disorders or in treatment with anticoagulant drugs;
* Patients suffering from dermatological diseases and connective tissue diseases;
* Patients suffering from other organic, psychiatric diseases or laboratory abnormalities could preclude participation or invalidate the study results;
* Inability to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
To use genetically encoded engineered proteins to obtain an inducible control of their activity in living human neurons preventing dendritic spines loss | 2 years
  The primary outcome measure will be the change in synaptic density (i.e., number of spines/micrometers) in living human neurons assessed using two-photon laser scanning microscopy.
To leverage genetically encoded engineered proteins to prevent alterations in the morphology of dendritic spines in living human neurons | 2 years
  Here the measure will be the change in dendritic spine morphology (evaluating the subtype of spines, i.e., thin, stubby, mushroom, etc.) in living human neurons assessed using two-photon laser scanning microscopy.
To use genetically encoded engineered proteins to obtain an inducible control of their activity in living human neurons promoting functional synaptic plasticity | 2 years
  The glutamatergic synaptic responses (i.e., AMPA receptor-mediated currents) will be measured in patch-clamp experiments in in living human neurons.
To use genetically encoded engineered proteins to obtain evaluate neuronal excitability in living human neurons | 2 years
  Neuronal excitability (i.e., number of action potentials recorded with depolarizing current injection) will be measured in patch-clamp experiments in in living human neurons.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy